CLINICAL TRIAL: NCT04651712
Title: The Effect of a Point-of-care Sputum Specimen Assay on Antibiotic Treatment of Patients Admitted Acutely With Suspected Pneumonia: A Multicenter Randomized Controlled Trial
Brief Title: The Effect of a Point-of-care Sputum Specimen Assay at the Emergency Department for Patients Suspected of Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHS-ED-11c-2020
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pneumonia, Bacterial
Keywords: Emergency department; Antibiotics; Sputum
MeSH Terms: conditions — Pneumonia, Bacterial; Emergencies

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be blinded, and the investigator will be blinded to POC-PCR results, data management and analysis, but not allocation. Outcome assessors will not be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): A treating physician must perform a clinical assessment within half an hour of patient arrival. This assessment includes the decision whether the patient is suspected of having pneumonia and if this is the case, a sputum specimen and chest x-ray will be ordered. Patients with suspected pneumonia who can deliver a sputum specimen will be randomly allocated with a 1:1 computer-generated randomization schedule with permuting blocks in relation to optimal therapeutical intervention strategy. All standard care sputum samples will be cultured and analysed according to the sites' standard procedures. Under standard care, the treating physician alone decides on the optimal therapeutical intervention.
- POC-PCR analysis supplied with a recommended action list developed by a microbiologist (Active Comparator): Along with standard analyses, the specimens will be analysed with POC-PCR and the treating physician will receive an action-list with the results from POC-PCR.
  Interventions: Diagnostic Test: POC-PCR

INTERVENTIONS:
Diagnostic Test: POC-PCR — The result of the POC-PCR will be presented by the study assistant to the treating physician within four hours upon admission. The treating physician will along with the result receive a recommended action list, developed by microbiologists.
  Arms: POC-PCR analysis supplied with a recommended action list developed by a microbiologist

SUMMARY:
Antibiotic resistance has been identified by the WHO as one of the biggest threats to the health of the world population. In Denmark, there has been an increasing focus on optimizing antibiotic consumption in recent years, but despite significant efforts, total consumption has increased in the hospital sector, especially regarding consumption and in the use of broad-spectrum antibiotics. Currently, a pneumonia diagnosis is primarily based on clinical symptoms such as cough, shortness of breath, chest pain, fever and sputum production, combined with X-ray of the lungs, relevant blood tests and microbiological analysis of sputum samples. X-ray is however an imprecise diagnostic tool, and sputum assays responses are available after 2 days. Sputum can be cultivated to determine the bacterial agent. However, the sputum samples are often of poor quality and many patients cannot deliver a sample. A recently published Danish study shows, that only half of the patients at the ED have sputum samples collected for culturing and none of them had the antibiotic treatment adjusted based on the microbiological results of the sputum.

This study's hypothesis is that point-of-care-polymerase chain reaction (POC-PCR) is superior to standard care on the prescription of targeted pneumonia treatment.

DETAILED DESCRIPTION:
The diagnosis of pneumonia is challenged by nonspecific symptoms, uncertain diagnostic methods, poor prognostic tools and waiting time for test results up to several days. A patient's length of stay in a Danish Emergency Department rarely exceeds 48 hours. Within this period the patient is examined, treated and discharged either home or to another department. Therefore, rapid molecular detection of respiratory pathogens is needed to add value to the management of the diagnostics of pneumonia and could reduce the initial use of antibiotics. Molecular diagnostic tests based on polymerase chain reaction (PCR) assays generate high sensitive analyses in one hour from specimen collection. The Biofire® FilmArray® Pneumonia Panel plus (Biomérieux) can identify 18 bacterial agents including 3 atypical pathogens 9 viruses and 7 antimicrobial resistance genes. This point-of-care (POC) test is promising, as bacterial pathogens often coexist with viruses or are identified with mixed infections. However, the high specificity of molecular diagnostics can challenge the interpretation of clinically significant agents and demands interpretation by highly qualified specialists. Therefore, the POC-PCR combined with advice from a microbiologist has the potential to optimize therapeutic regimens and reduce prescriptions of inappropriate broad-spectrum antibiotics in the initial management of pneumonia.

This study aims to

* investigate how effective the addition of POC-PCR analysis of sputum is to the diagnostic set-up for community-acquired pneumonia on antibiotic prescription at 4 hours after admission without consequent adverse advents
* to identify the effect of POC-PCR on prescribed antibiotic treatment 48 hours after admission and 24 hours after discharge
* to investigate the agreement between POC-PCR and sputum culture on microbiological analysis

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patients suspected of pneumonia by the attending physician and with at least one of the following symptoms: dyspnea, cough, expectoration, chest tightness or fever and indication for chest x-ray

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Antibiotic treatment at 4-hour plan | 4 hours after admission
  The primary outcome is to determine the effectiveness of POC-PCR sputum analysis on antibiotic prescription, the treatment will either be registered as targeted or non-targeted antibiotic treatment at four hours after admission. This is a binary outcome.

SECONDARY OUTCOMES:
Intensive care unit (ICU) treatment | within 60 days from admission to the emergency department
  Transfer to the intensive care unit will be recorded during the current hospitalization as a binary variable (transferred/not-transferred)
Length of hospital stay | within 60 days from current admission to the emergency department
  Defined as the time (in days) spent in hospital during the current admission. Measured in days from admission to hospital discharge. Discharge date minus admission date.
30-days mortality | 30 days from the admission to the emergency department
  Mortality within 30 days from admission to the Emergency Department
Readmission | within 30 days from the discharge to the hospital
  If a subject is admitted over a 30 day period after the current hospitalization discharge measured as a binary outcome Re-admissions/not re-admissions.
In-hospital mortality | within 60 days from admission to the emergency department
  Patient mortality during the current hospitalization. Binary outcome - Died/ Not died
Antibiotic treatment at 48 hour | 48 hours after admission
  The treatment will either be registered as targeted or non-targeted antibiotic treatment 48 hours after admission. This is a binary outcome.
Antibiotic treatment at discharge from hospital | 24 hours after hospital discharge
  The treatment will either be registered as a targeted or non-targeted antibiotic treatment after the patient is discharged from the hospital. This is a binary outcome.
Bacterial agents and viruses from the microbiological results | Within the first 7 days from specimen collection
  The bacterial agents and viruses from the Biofire® FilmArray® Pneumonia Panel plus (Biomérieux) and standard sputum culture for the two microbiological analysis will be presented as descriptive statistics.

OTHER OUTCOMES:
CURB-65 score for pneumonia severity | within 4 hours from admission
  Confusion of new onset, Blood Urea nitrogen greater than 7 mmol/L (19 mg/dL), respiratory rate of 30 breaths per minute or greater, blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less and age 65 or older
Pneumonia severity index (PSI) | within 4 hours from admission
  Risk classes to predict the severity of pneumonia. Scores are given based on demographics, comorbidity, clinical measurements and physical Exam Findings (<70 = Risk Class II, 71-90 = Risk Class III, 91-130 = Risk Class IV, >130 = Risk Class V)
Number of clostridium infections | measured 40 days after discharge from the emergency department
  Identify through patient records if the patient was infected with clostridium difficille, binary outcome yes/no
Procalcitonin (PCT), Soluble Urokinase Plasminogen Activator Receptor (suPAR), YKL-40 and Krebs von den Lungen (KL-6) | results within 4 hour from admission
  Measurement of serum PCT and suPAR are collected in connection to routine blood tests within 1 hour from admission
90 days mortality | Within 90 days from admission to emergency department
  binary

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, MD PhD, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skjot-Arkil H, Mogensen CB, Lassen AT, Johansen IS, Chen M, Petersen P, Andersen KV, Ellermann-Eriksen S, Moller JM, Ludwig M, Fuglsang-Damgaard D, Nielsen FE, Petersen DB, Jensen US, Rosenvinge FS. Carrier prevalence and risk factors for colonisation of multiresistant bacteria in Danish emergency departments: a cross-sectional survey. BMJ Open. 2019 Jun 27;9(6):e029000. doi: 10.1136/bmjopen-2019-029000. PMID 31253624
- [Background] Sogaard M, Nielsen RB, Schonheyder HC, Norgaard M, Thomsen RW. Nationwide trends in pneumonia hospitalization rates and mortality, Denmark 1997-2011. Respir Med. 2014 Aug;108(8):1214-22. doi: 10.1016/j.rmed.2014.05.004. Epub 2014 May 20. PMID 24898129
- [Background] Welte T, Torres A, Nathwani D. Clinical and economic burden of community-acquired pneumonia among adults in Europe. Thorax. 2012 Jan;67(1):71-9. doi: 10.1136/thx.2009.129502. Epub 2010 Aug 20. PMID 20729232
- [Background] van der Eerden MM, Vlaspolder F, de Graaff CS, Groot T, Bronsveld W, Jansen HM, Boersma WG. Comparison between pathogen directed antibiotic treatment and empirical broad spectrum antibiotic treatment in patients with community acquired pneumonia: a prospective randomised study. Thorax. 2005 Aug;60(8):672-8. doi: 10.1136/thx.2004.030411. PMID 16061709
- [Background] Becerra MB, Becerra BJ, Banta JE, Safdar N. Impact of Clostridium difficile infection among pneumonia and urinary tract infection hospitalizations: an analysis of the Nationwide Inpatient Sample. BMC Infect Dis. 2015 Jul 1;15:254. doi: 10.1186/s12879-015-0925-9. PMID 26126606
- [Background] Ewig S, Schlochtermeier M, Goke N, Niederman MS. Applying sputum as a diagnostic tool in pneumonia: limited yield, minimal impact on treatment decisions. Chest. 2002 May;121(5):1486-92. doi: 10.1378/chest.121.5.1486. PMID 12006433
- [Background] Roson B, Carratala J, Verdaguer R, Dorca J, Manresa F, Gudiol F. Prospective study of the usefulness of sputum Gram stain in the initial approach to community-acquired pneumonia requiring hospitalization. Clin Infect Dis. 2000 Oct;31(4):869-74. doi: 10.1086/318151. Epub 2000 Oct 12. PMID 11049763
- [Background] Hadfield J, Bennett L. Determining best outcomes from community-acquired pneumonia and how to achieve them. Respirology. 2018 Feb;23(2):138-147. doi: 10.1111/resp.13218. Epub 2017 Nov 17. PMID 29150897
- [Derived] Cartuliares MB, Rosenvinge FS, Mogensen CB, Skovsted TA, Andersen SL, Ostergaard C, Pedersen AK, Skjot-Arkil H. Evaluation of point-of-care multiplex polymerase chain reaction in guiding antibiotic treatment of patients acutely admitted with suspected community-acquired pneumonia in Denmark: A multicentre randomised controlled trial. PLoS Med. 2023 Nov 28;20(11):e1004314. doi: 10.1371/journal.pmed.1004314. eCollection 2023 Nov. PMID 38015833
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497